CLINICAL TRIAL: NCT02640677
Title: 4CMenB Pregnancy Registry: an Observational Study of the Safety of 4CMenB Exposure in Pregnant Women and Their Offspring.
Brief Title: Safety of 4CMenB Exposure During Pregnancy
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 205533; V72_82OB (Other: Novartis); EUPAS 12183 (Registry Identifier: EU PAS)
Record Dates: First submitted 2015-12-21; First posted 2015-12-29 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Infections, Meningococcal
MeSH Terms: conditions — Meningococcal Infections | interventions — 4CMenB vaccine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pregnant women exposed to 4CMenB: Pregnant women within the United States (U.S) who received at least 1 dose of 4CMenB vaccine within 30 days prior to Last Menstrual Period (LMP) or at any time during pregnancy
  Interventions: Biological: 4CMenB

INTERVENTIONS:
Biological: 4CMenB — This study is strictly observational; Administration of BEXSERO, the schedule of office visits and all treatment regimens will be determined by the treating health care provider in the context of routine clinical care.

SUMMARY:
4CMenB was approved by the Food and Drug Administration (FDA) in the United States in January 2015 for people aged 10 through 25 years of age. 4CMenB should be used during pregnancy only if clearly needed and sometimes, inadvertent exposure during pregnancy may also occur - before the woman knows she is pregnant, for example. The objective of this study is to evaluate the safety of 4CMenB during pregnancy and to help us learn more about the health of women who have been vaccinated with 4CMenB within 30 days prior to their last menstrual period (LMP) or at any time during pregnancy, and the health of their infants. Pregnant women within the US who received at least 1 dose 4CMenB vaccine within 30 days prior to their last menstrual period or at any time during pregnancy are eligible to participate. A woman may self-enroll in the registry by calling the pregnancy registry telephone number directly or their healthcare provider (HCP) can, with their consent, enroll them on their behalf. Alternatively HCPs may report anonymous data on pregnancy exposures and outcomes occurring within their network/health maintenance organization (HMO). The health of the woman and her infant will be followed up until the end of the pregnancy.

ELIGIBILITY:
Inclusion Criteria:

Any pregnant women within the US who received at least 1 dose 4CMenB vaccine within 30 days prior to LMP or at any time during pregnancy where:

* Sufficient evidence to confirm that exposure to a meningococcal B vaccine (confirmed or possible 4CMenB exposure) occurred within 30 days prior to LMP or at any time during pregnancy
* Sufficient information to determine whether the pregnancy is prospectively or retrospectively registered (i.e., whether the outcome of pregnancy was known at the time of first contact with the registry)
* Date the pregnancy exposure is registered
* Full reporter (i.e., HCP) contact information to allow for follow-up (name, address, etc.)

Exclusion Criteria:

Pregnant women vaccinated with a different brand of Meningococcal B vaccine will not be included. (Of note: In the event that it cannot be ascertained to which meningococcal B vaccine the woman was exposed, an unknown exposure cohort will be established and analyzed separately).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include pregnant women within the US who received at least 1 dose 4CMenB vaccine within 30 days prior to LMP or at any time during pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2016-01-31 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wilmington, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At the end of recruitment of this pregnancy registry for Bexsero, there were only 2 registrations. Of these,1 subject withdrew the consent and the other subject did not return for a follow up, hence considered as lost to follow up. Therefore, no pregnancy outcome data are available for this study.
Groups:
- Pregnant Women Exposed to 4CMenB: Pregnant women within the United States (US) who received at least 1 dose of 4CMenB vaccine within 30 days prior to Last Menstrual Period (LMP) or at any time during pregnancy
Period: Overall Study
Arm/Group | Pregnant Women Exposed to 4CMenB
Started | 2
Completed | 0
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pregnant Women Exposed to 4CMenB
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic ethinicity | 2

OUTCOME MEASURES:

1. Primary Outcome: Major Congenital Malformation (MCM)
Time Frame: At registry enrollment
Population: Data was not collected for this outcome measure as the enrolled participants did not complete the study
Arm/Group | Pregnant Women Exposed to 4CMenB
Number analyzed (Participants) | 0

2. Primary Outcome: Preterm Birth
Time Frame: At registry enrollment
Population: Data was not collected for this outcome measure as the enrolled participants did not complete the study
Arm/Group | Pregnant Women Exposed to 4CMenB
Number analyzed (Participants) | 0

3. Primary Outcome: Low Birth Weight (LBW)
Time Frame: At registry enrollment
Population: Data was not collected for this outcome measure as the enrolled participants did not complete the study
Arm/Group | Pregnant Women Exposed to 4CMenB
Number analyzed (Participants) | 0

4. Secondary Outcome: Spontaneous Abortions and Still Births
Time Frame: At registry enrollment
Population: Data was not collected as the enrolled participants did not complete the study
Arm/Group | Pregnant Women Exposed to 4CMenB
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Safety data was not collected from any participant in this study
Description: Safety data was not collected from any participant in this study
Arm/Group | Pregnant Women Exposed to 4CMenB
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT02640677/Prot_SAP_000.pdf